CLINICAL TRIAL: NCT07292805
Title: Bronchial Thermoplasty (BT) for Severe Asthma in the Biologic Era: a Randomized Controlled Trial (BOOSTER Trial)
Brief Title: Bronchial Thermoplasty for Adults With Severe Asthma in the Biologic Era
Acronym: BOOSTER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Peter I. Bonta, MD PhD, MD PhD, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL85642.018.23
Record Dates: First submitted 2025-01-22; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Asthma Exacerbations; Severe Asthma; Bronchial Thermoplasty
Keywords: bronchial thermoplasty; asthma; severe asthma; asthma exacerbations
MeSH Terms: conditions — Asthma | interventions — Bronchial Thermoplasty

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Usual care for patient with severe asthma
- Intervention - Bronchial thermoplasty (Active Comparator): Intervention with bronchial thermoplasty
  Interventions: Procedure: Bronchial thermoplasty

INTERVENTIONS:
Procedure: Bronchial thermoplasty — Bronchial thermoplasty will be performed according to prior SOP's, in three sessions. First session RLL, second session LLL, third session RUL/LUL
  Arms: Intervention - Bronchial thermoplasty

SUMMARY:
Rationale: For patients with severe asthma that remain uncontrolled with exacerbations despite biologics or patients who are not eligible for biologics, there is no reimbursed treatment other than pulmonary rehabilitation in the Netherlands. Pulmonary rehabilitation is known to have a limited effect for a limited amount of time. Bronchial thermoplasty or bronchial ablation (BT) is a non-pharmacological treatment for asthma aiming to restore abnormal airway function by using an endobronchial approach. Previous RCT's reported efficacy on exacerbations and asthma related quality of life (AQLQ), but were performed before large availability of biologic treatments. Although a single BT treatment is not without costs, these costs seem to outweigh the costs that can be saved by the long-term (>5 years) lowering effect of BT on the frequency of exacerbations and hospitalizations and omitting long term use of trials and switches of biologics. Therefore, the investigators hypothesize that BT, in the era of biologics, is superior (in terms of exacerbations and quality of life) over standard care and cost-effective in patients whose asthma remains uncontrolled despite optimal anti-inflammatory treatments including biologics, and the investigators propose to test this hypothesis in a RCT.

Objective: To investigate the impact of BT as compared to standard of care in severe asthma patients that remain uncontrolled despite standard treatment including adequate doses of inhaled preventer therapies with or without biologics on:

1. rate of exacerbations
2. asthma related quality of life (AQLQ)
3. 1-year and 5-year cost-effectiveness and cost utility Study design: Investigator-initiated randomized, multicenter, parallel-group interventional RCT of severe asthma patients undergoing either BT (active arm) or standard care (control arm).

Study population: Adult, uncontrolled severe asthma patients despite optimal medical therapy including one or more trials of treatment with a biologic or ineligible for biologic treatment AND 2 or more severe asthma exacerbations in the previous year AND FEV1 ≥ 50% predicted.

Intervention: BT (active arm) versus standard care (control arm). Main study parameters/endpoints: The primary endpoint of this study is the between group difference in severe exacerbation rate after 12 months of follow-up. The main secondary endpoints are between group differences after 12 months of follow-up and within group differences before and after intervention or standard care. Parameters that will be explored are: AQLQ (minimal clinically important difference >0.5), ACQ (minimal clinically important difference >0.5), exacerbation rate (before and after BT) and hospitalizations (rate and % subjects).

DETAILED DESCRIPTION:
An estimated 3.6% of asthma patients suffer from severe asthma with frequent exacerbations, decreased quality of life and excessive health care utilisation. Clinical guidelines recommend treatment with high-dose inhaled corticosteroids (ICS) and bronchodilators in these patients. If their asthma remains uncontrolled (or if they require continuous oral corticosteroids (OCS)), add-on treatment with biologics, macrolides, pulmonary rehabilitation or bronchial thermoplasty (BT) should be considered. Treatment with biologics have rapidly emerged and includes anti-IgE (Immunoglobulin E; Omalizumab), anti-interleukin (IL)-5 (Reslizumab, Benralizumab, Mepolizumab), or anti-IL-4 (Dupilumab). Although the currently available biologics are effective in many patients with severe asthma with type-2 inflammation, a substantial proportion do not respond to biologics, or only respond partially. In addition, not all severe asthma patients have a phenotype that is eligible for biologic treatment. Because there are currently no wellestablished treatments available for patients with uncontrolled asthma despite or ineligible for biologic treatment, these patients have a high burden of disease with impaired lung function, frequent or persistent use of OCS (with high risk of long-term adverse effects), and high medical and societal costs due to exacerbations resulting in frequent hospital visits, admissions and sick leave. There is an urgent need for effective therapies in these patients.

BT is a non-pharmacological treatment for asthma aiming to permanently restore abnormal airway function by using an endobronchial approach. During this procedure, which is performed by a pulmonologist, radiofrequent energy at 65°C is delivered locally to the airways, with the patient under deep sedation or general anesthesia, in three sessions with three week intervals. In the first session, the right lower lobe is treated, followed by the left lower lobe in the second session, and both upper lobes in the last session. In contrast to corticosteroids and biologics, which act on inflammation, BT modifies airway remodelling, which is one of the hallmarks of pathophysiology in asthma. In mechanistic studies, BT had multilevel impact on airway remodelling with a reduction in airway smooth muscle, extra cellular matrix and innervation, and a healthier state of the epithelium, providing a complementary effect to corticosteroids and biologics. Although patients may experience a transient increase in respiratory symptoms in-between BT-sessions, multiple randomized clinical trials (RCTs) and post-FDA (Federal Drug Administration) approval monitoring registries (and meta-analyses of the results of these studies) have shown that BT is safe and improves clinically relevant asthma outcomes (e.g. exacerbations and quality of life) for years afterwards. Based on this, guidelines including GINA (Global Initiative for Asthma), NICE (National Institute for Health and Care Excellence; and NVALT (Dutch Pulmonology Society) recommend that BT should be considered as a treatment for severe uncontrolled asthma. These recommendations have resulted in the conditional re-imbursement of BT in several countries (e.g. UK, France, Spain, Germany, Italy, US, Japan, China and Australia).

In 2019, on behalf of the NVALT, the investigators applied for reimbursement/insurance of BT in severe asthma in the Netherlands.

Although judged as promising ('veelbelovend'), the request was denied by an ad-hoc committee of 'Zorgverzekeraars Nederland', mainly advocated by inconsistency in primary endpoints and patient populations across the three available RCTs, and because most of the data had been obtained before the widespread use of biologics.

Due to these deficiencies, it is currently under debate wheter or not BT is superior over standard care in patients with severe uncontrolled asthma despite or ineligible for biologic treatment. Since 2014, our group has performed the TASMA study, a RCT comparing immediate BT with delayed BT in severe asthma patients. On the primary endpoint, a significant reduction in airway smooth muscle was observed. Results on secondary endpoints mirrored those of earlier RCTs in terms of clinical efficacy (reduction in exacerbations and improvement in ACQ (Asthma Control Questionnaire) and AQLQ (Asthma Quality of Life Questionnaire)) and safety. In addition, in line with others, the investigators showed that BT was effective even in patients taking high doses of anti-inflammatory treatments, including OCS and biologics. This confirms that BT is a promising treatment for patients with severe asthma who do not or cannot benefit from biologics. For patients with severe asthma that remain uncontrolled with exacerbations despite biologics or patients who are not eligible for biologics, there is no approved treatment other than pulmonary rehabilitation, which is known to have a limited effect for a limited amount of time. Although a single BT treatment is not without costs, these costs far outweigh the costs that can be saved by the long-term (>5 years) lowering effect of BT on the frequency of exacerbations and hospitalizations and omitting long term use or trials and switches of biologics. Therefore, the investigators hypothesize that BT is superior (in terms of exacerbations and quality of life) over standard care and cost-effective in patients whose asthma remains uncontrolled despite optimal anti-inflammatory treatments including biologics, and the investigatorspropose to test this hypothesis in a RCT.

ELIGIBILITY:
Inclusion Criteria:

* adult (>18 years)
* severe uncontrolled asthma (defined as ACQ above 1.5) despite optimal medical therapy (GINA treatment step 5; alternative diseases excluded, therapy compliance and adequate inhalation technique confirmed)
* 1 or more trials of treatment with a biologic or ineligible for biologic treatment
* 2 or more severe asthma exacerbations in the previous year (defined as the need for a course of OCS or doubling dose of maintenance OCS for at least 3 consecutive days)
* FEV1 ≥ 50% predicted after 400μg inhaled salbutamol or equivalent

Exclusion Criteria:

* chronic OCS therapy at a dose >20 mg/day prednisone equivalent
* 1 or more ICU admission for mechanical or endotracheal intubation for
* asthma in the previous year.
* anti-coagulation therapy that cannot be stopped temporarily
* pregnancy
* body mass index ≥35
* current or ex-smokers with >20 pack years
* DLCOc <70%
* Subject has a known sensitivity to medications required to perform bronchoscopy
* Subject is using immunosuppressant therapy other than oral steroid therapy that impact on BT
* Subject has bleeding diathesis, platelet dysfunction, thrombocytopenia with platelet count less than 100,000/mm2 or known coagulopathy
* Comorbidities that are a contra-indication for BT such as severe heart failure and other respiratory diseases including bronchiectasis, interstitial lung disease, emphy-sema, cystic fibrosis, mechanical upper airway obstruction, Churg-Strauss syndrome, and allergic bronchopulmonary aspergillosis (ABPA)
* Subject uses an internal or external pacemaker or cardiac defibrillator..

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Exacerbation | 12 months
  severe exacerbation rate after 12 months of follow-up

SECONDARY OUTCOMES:
Asthma related quality of life | 12 months
  Asthma related quality of life:
  AQLQ questionnaire (minimal clinically important difference >0.5)
Symptom burden | 12 months
  Asthma related symptom burden Measured by ACQ questionnaire (minimal clinically important difference >0.5)
Emergency department visits | 12 months
  Number of emergency department visits 12 months after treatment/start of follow up (rate and % subjects)
Hospitalizations | 12 months
  Number of hospitalizations due to asthma exacerbations in 12 months following treatment/start follow-up (rate and % subjects)
Maintenance OCS use | 12 months
  If patients is using maintenance oral corticosteroids 12 months after treatment/starty follow-up (Number of patients and difference (%) between baseline and 12 months follow-up.
Biological use | 12 months
  The number of patients that use a biologic for asthma at 12 months after treatment/start follow-up, as compared to baseline and between groups (number and % subjects)
Treatment related adverse events | 12 months
  The number and severeity of adverse events in the group of subjects that are treated with bronchial thermoplasty and are followed-up

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - amsterdam UMC, Amsterdam
  - UMCG, Groningen

IPD SHARING:
Plan to Share IPD: Yes
all IPD collected throughout the trial
Supporting Information: Study Protocol